CLINICAL TRIAL: NCT02911194
Title: A1 Beta Casein Free Milk (a2 Milk) for Autism and Attention-deficit Hyperactivity Disorder
Brief Title: a2 Milk for Autism and Attention-deficit Hyperactivity Disorder (ADHD)
Acronym: A2MT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: ESPA Research (Unknown); a2 Milk Company Ltd. (Industry)
Responsible Party: Principal Investigator, John Lodge, Doctor, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SUB017_Lodge_031115
Record Dates: First submitted 2016-07-22; First posted 2016-09-22 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Autism; Attention Deficit Hyperactivity Disorder; Autism Spectrum Disorder
MeSH Terms: conditions — Autistic Disorder; Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): a2 milk intervention period
  Interventions: Dietary Supplement: a2 milk
- Control (Placebo Comparator): a1 containing milk (normal) intervention period
  Interventions: Dietary Supplement: a1 containing milk

INTERVENTIONS:
Dietary Supplement: a2 milk — replace all milk with a2 milk
  Arms: Treatment
Dietary Supplement: a1 containing milk — use a1 containing milk
  Arms: Control

SUMMARY:
Under double-blind, placebo-controlled, cross-over conditions, the short-term effects of use of A1 beta casein free milk (a2 milk) and milk containing A1 beta casein will be compared in a sample of pre-pubescent boys diagnosed with an autism spectrum disorder (ASD) with concurrent features of attention-deficit hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
Previous preliminary research studies have suggested that a diet devoid of milk and dairy products might be useful for some people on the autism spectrum in reducing certain types of behaviours or other symptoms that can affect quality of life. Aggravation of some of the symptoms of autism has been suggested to be linked to some of the constituents of milk, in particular a natural breakdown product of the milk protein called beta-casomorphin 1-7 (BC 1-7 or BCM-7) found in the majority of mammalian dairy products. A dairy-free diet (casein-free diet) can however be a difficult diet to follow and may increase the risk that certain nutrients are missing from the diet.

Anecdotal evidence suggests that different types of milk from different breeds of cattle (cows) may not carry the same biological effects for some on the autism spectrum. Milk typically found in supermarkets naturally contains BC1-7 as a function of the type of cows producing the milk and the protein it contains (A1 variant of the beta casein protein).

The investigators are aiming to test whether a particular type of milk (A1 beta casein free milk also called a2 Milk™) might be able to replace a casein-free diet for children on the autism spectrum also presenting with attention-deficit hyperactivity disorder (ADHD) type symptoms. The investigators will be looking at the potential effects of A1 beta casein free milk on behaviour and various biological processes going on in the body. The source of A1 beta casein free milk will be commercially available a2 Milk™ branded milk that is directly comparable to regular supermarket bought milk with the exception of the beta casein component and is already available to buy.

In this double-blind, randomised, placebo-controlled trial, the effects of milk free of A1 beta casein (a branded milk called a2 milk™) and milk containing A1 beta casein will be compared in a sample of pre-pubescent children diagnosed with an autism spectrum disorder with concurrent features of attention-deficit hyperactivity disorder (ADHD). Forty children based in North East England will be initially recruited; all possessing communicative speech and language. A baseline assessment will be conducted to include behavioural, psychometric and health-related parameters. Following random allocation, participants will be assigned to group A or group B and given A1 milk or a2 Milk™ initially for a period of 4 weeks. At this point, baseline assessment measures will be repeated. Milk types will be crossed for groups for a further 4 weeks. At study endpoint, baseline assessment measures will be repeated again. Data derived from the study will be analysed and outcomes reported in peer-review format. During the course of the study, all other forms of dairy product consumption (cheese, yogurts, etc) will be excluded from the diet of all participants irrespective of their treatment allocation.

Data from supervised baseline, midpoint and endpoint psychometric and behavioural assessments will be made and stored via a secure survey website accessed via tablets supplied to all participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism spectrum disorder (autism, Asperger syndrome, Autism Spectrum Disorder)
* Diagnosis or fulfilling the diagnostic criteria for / presenting with the symptoms of attention-deficit hyperactivity disorder (ADHD)
* Regular milk drinker
* Functional use of spoken language (for ability to self-report)
* Access to internet connection (WiFi)

Exclusion Criteria:

* Undergoing current medical treatment (and an inpatient at a state hospital)
* Current or past 3 month use of a gluten- and/or casein-free diet
* Co-morbid diagnoses of Fragile-X syndrome, epilepsy or tuberous sclerosis
* Indications or diagnosis of cows milk protein allergy (IgE)

Ages: 5 Years to 10 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-09; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Change in Childhood Autism Rating Scale (CARS2-HF) Value during intervention | Baseline to Week 4 to Week 8
  Difference in CARS raw scores and severity group between baseline and 4 weeks and 8 weeks.
Change in Conners' Rating Scale - Revised (L) value during intervention. | Baseline to Week 4 to Week 8
  Difference in Conners' raw scores and totalled scores between baseline and 4 weeks and 8 weeks

SECONDARY OUTCOMES:
Amino acid analysis of urine samples by mass spectroscopy. | Baseline to Week 4 to Week 8
  Analysis of urine samples via non-targeted and targeted liquid chromatography mass spectrometry analysis. The targeted compounds to be measured include urinary metabolites of intestinal bacterial species (specifically related to the aromatic amino acids, tryptophan, tyrosine and phenylalanine) and urinary concentrations of compounds related to the methionine cycle (including methionine, homocysteine, cystathione and cysteine).
Metabolomic analysis of blood spot samples by mass spectroscopy. | Baseline to Week 4 to Week 8
  Where blood spot samples are/can be provided by participants, non-targeted and targeted liquid chromatography mass spectrometry analysis will be undertaken. The targeted compounds to be measured include various amino acids including the aromatic amino acids and the branched chain amino acids. Blood spot concentrations of compounds related to the methionine cycle (including methionine, homocysteine, cystathione and cysteine) will also be examined.
Changes to the gut microbiome profile. | Baseline to Week 4 to Week 8
  Gene sequencing of stool samples to characterise the gut microbiome measured by operational taxonomic units (OTUs) of individual bacterial species.
Changes to stool appearance measured using the Bristol Stool Chart. | Baseline to Week 4 to Week 8
  At time of stool sample collection, the presentation of the stool will be recorded using the Bristol Stool Chart.

CONTACTS AND LOCATIONS:
Overall Officials: John K Lodge, PhD, Principal Investigator — Northumbria University
Locations (1):
- ESPA Research, Sunderland, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Group data will be available upon request

REFERENCES:
- [Background] Whiteley P. Nutritional management of (some) autism: a case for gluten- and casein-free diets? Proc Nutr Soc. 2015 Aug;74(3):202-7. doi: 10.1017/S0029665114001475. Epub 2014 Oct 14. PMID 25311313
- [Background] Pedersen L, Parlar S, Kvist K, Whiteley P, Shattock P. Data mining the ScanBrit study of a gluten- and casein-free dietary intervention for children with autism spectrum disorders: behavioural and psychometric measures of dietary response. Nutr Neurosci. 2014 Sep;17(5):207-13. doi: 10.1179/1476830513Y.0000000082. Epub 2013 Nov 26. PMID 24075141
- [Background] Whiteley P, Shattock P, Knivsberg AM, Seim A, Reichelt KL, Todd L, Carr K, Hooper M. Gluten- and casein-free dietary intervention for autism spectrum conditions. Front Hum Neurosci. 2013 Jan 4;6:344. doi: 10.3389/fnhum.2012.00344. eCollection 2012. PMID 23316152
- [Background] Whiteley P, Haracopos D, Knivsberg AM, Reichelt KL, Parlar S, Jacobsen J, Seim A, Pedersen L, Schondel M, Shattock P. The ScanBrit randomised, controlled, single-blind study of a gluten- and casein-free dietary intervention for children with autism spectrum disorders. Nutr Neurosci. 2010 Apr;13(2):87-100. doi: 10.1179/147683010X12611460763922. PMID 20406576
- [Background] Jianqin S, Leiming X, Lu X, Yelland GW, Ni J, Clarke AJ. Effects of milk containing only A2 beta casein versus milk containing both A1 and A2 beta casein proteins on gastrointestinal physiology, symptoms of discomfort, and cognitive behavior of people with self-reported intolerance to traditional cows' milk. Nutr J. 2016 Apr 2;15:35. doi: 10.1186/s12937-016-0147-z. PMID 27039383
- [Background] Ho S, Woodford K, Kukuljan S, Pal S. Comparative effects of A1 versus A2 beta-casein on gastrointestinal measures: a blinded randomised cross-over pilot study. Eur J Clin Nutr. 2014 Sep;68(9):994-1000. doi: 10.1038/ejcn.2014.127. Epub 2014 Jul 2. PMID 24986816
- [Background] Trivedi MS, Shah JS, Al-Mughairy S, Hodgson NW, Simms B, Trooskens GA, Van Criekinge W, Deth RC. Food-derived opioid peptides inhibit cysteine uptake with redox and epigenetic consequences. J Nutr Biochem. 2014 Oct;25(10):1011-8. doi: 10.1016/j.jnutbio.2014.05.004. Epub 2014 Jun 6. PMID 25018147
- See also: ESPA Research website — http://www.espa-research.org.uk